CLINICAL TRIAL: NCT04600492
Title: The Effect of Riociguat for Peak Cardiac Index on Cardiopulmonary Exercise Test in CTEPH Patients After Normalization of Pulmonary Artery Pressure by Combination Treatment of Riociguat and Balloon Pulmonary Angioplasty
Brief Title: THERAPY-HYBRID-BPA Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Hospital Organization Okayama Medical Center (Other)
Collaborators: Bayer Yakuhin, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Riociguat-CTEPH
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Hypertension, Pulmonary
Keywords: Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — riociguat

STUDY DESIGN:
Intervention Model Description: A double-blind, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: A double-blind, placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Active drug group Riociguat (Active Comparator): Riociguat 0.5mg、1.0mg、2.5mg
  Interventions: Drug: Riociguat Oral Tablet
- Placebo group (Placebo Comparator): Placebo 0.5mg、1.0mg、2.5mg
  Interventions: Drug: Riociguat Oral Tablet

INTERVENTIONS:
Drug: Riociguat Oral Tablet — Take any dose of Riociguat from 0.5mg to 2.5mg, or placebo

SUMMARY:
Riociguat could improve the exercise capacity and residual symptoms in patients with chronic thromboembolic pulmonary hypertension (CTEPH) even after normalization of pulmonary arterial pressure by balloon pulmonary angioplasty (BPA). This randomized controlled trial study aimed to clarify whether the improvement of peak cardiac index (CI) during exercise maintains or not between the riociguat continued group and the riociguat discontinued group.

DETAILED DESCRIPTION:
CTEPH is a disease that causes progressive pulmonary hypertension due to stenoses or occlusions in the pulmonary artery due to an organized thrombus. And this is a disease that results in right heart failure and death unless early diagnosis and appropriate treatment are performed. Pulmonary endarterectomy (PEA), which surgically removes the intimal thrombus, has been established as the treatment of choice for CTEPH. In the AHA/ACC guideline and ESC guideline, PEA for CTEPH is class IC (1). In 2014, a soluble guanylate cyclase stimulant (generic name: riociguat), which is one of the therapeutic agents for pulmonary hypertension, was approved for patients with CTEPH who are ineligible for PEA, and residual pulmonary hypertension after PEA (2). In addition, it has been reported that BPA, which is a catheter interventional treatment, is also effective to improve hemodynamics in inoperable patients with CTEPH (3, 4). However, some patients have residual symptoms such as dyspnea on exertion even after normalization in hemodynamics by BPA. A randomized control study should be done to confirm the necessary of continuation of riociguat for such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet CTEPH diagnostic criteria (complying with 2017 Japanese Cardiovascular Society Guidelines diagnostic criteria)
2. Patients with diagnosed as a contraindication of pulmonary endarterectomy by an experienced surgeon in the central diagnosis
3. Patients who were adjusted to reach the appropriate dose of riociguat within 8 weeks and were able to continue riociguat thereafter
4. Patients who underwent BPA once or more after the dose adjustment of riociguat
5. Patients who have been able to continue taking the same dose of riociguat for more than 3 months
6. Patients who can obtain written informed consent from the patients and legal representatives
7. Patients with WHO functional class II or III at the time of the allocation
8. Over the age of 18 and under 85 at the time of obtaining informed consent
9. Patients with the resting CI value of less than 3.0 L/min/m2 in the right heart catheterization test immediately before the allocation
10. Patients with the mean pulmonary artery pressure less than 25 mmHg in a right heart catheterization test immediately before the allocation

Exclusion Criteria:

1. Patients who are eligible for pulmonary endarterectomy (PEA)
2. Patients with pulmonary hypertension other than class 4 by NICE classification
3. Patients having difficulty in performing cardiopulmonary exercise test (CPET)
4. Patients with severe right heart failure requiring cardiotonic drugs
5. Patients with severe heart disease
6. Patients with severe liver damage
7. Patients with systolic blood pressure less than 90 mmHg at the screening
8. Patients with shunt disease
9. Patients with severe renal dysfunction (CCr < 15 mL/min) requiring hemodialysis
10. Patients with life expectancy less than 2 years
11. Being pregnant or lactating
12. Patients who are contraindicated for riociguat
13. Patients using other unlicensed drugs
14. Patients who used pulmonary vasodilators within 4 weeks after obtaining the informed consent of the right heart catheterization test.
15. Patients whom the investigator determines that the participation in this study is inappropriate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-10-16 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2025-01-28 (Estimated)

PRIMARY OUTCOMES:
Peak CI change | from baseline to 16 weeks
  Change in Peak CI during the cardiopulmonary exercise test (CPET)

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Ito, Study Director — National Hospital Organization Nagoya Medical Center
Locations (1):
- National Hospital Org anization Okayama Medical Center, Okayama, Japan

REFERENCES:
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Background] Ghofrani HA, D'Armini AM, Grimminger F, Hoeper MM, Jansa P, Kim NH, Mayer E, Simonneau G, Wilkins MR, Fritsch A, Neuser D, Weimann G, Wang C; CHEST-1 Study Group. Riociguat for the treatment of chronic thromboembolic pulmonary hypertension. N Engl J Med. 2013 Jul 25;369(4):319-29. doi: 10.1056/NEJMoa1209657. PMID 23883377
- [Background] Mizoguchi H, Ogawa A, Munemasa M, Mikouchi H, Ito H, Matsubara H. Refined balloon pulmonary angioplasty for inoperable patients with chronic thromboembolic pulmonary hypertension. Circ Cardiovasc Interv. 2012 Dec;5(6):748-55. doi: 10.1161/CIRCINTERVENTIONS.112.971077. Epub 2012 Nov 27. PMID 23192917
- [Background] Kataoka M, Inami T, Hayashida K, Shimura N, Ishiguro H, Abe T, Tamura Y, Ando M, Fukuda K, Yoshino H, Satoh T. Percutaneous transluminal pulmonary angioplasty for the treatment of chronic thromboembolic pulmonary hypertension. Circ Cardiovasc Interv. 2012 Dec;5(6):756-62. doi: 10.1161/CIRCINTERVENTIONS.112.971390. Epub 2012 Nov 6. PMID 23132237
- [Derived] Shimokawahara H, Nishizaki M, Inami T, Kubota K, Taniguchi Y, Miyagi A, Kikuchi H, Goda A, Miyanaga S, Hashimoto H, Saito AM, Sekimizu M, Matsubara H. Effect of riociguat on exercise following balloon pulmonary angioplasty in patients with inoperable chronic thromboembolic pulmonary hypertension in Japan (THERAPY-HYBRID-BPA): a multicentre, double-blind, randomised, controlled, phase 4 trial. Lancet Respir Med. 2025 Sep;13(9):789-799. doi: 10.1016/S2213-2600(25)00127-4. Epub 2025 Jul 23. PMID 40714010
- [Derived] Shimokawahara H, Inami T, Kubota K, Taniguchi Y, Hashimoto H, Saito AM, Sekimizu M, Matsubara H. Protocol for a multicentre, double-blind, randomised, placebo-controlled trial of riociguat on peak cardiac index during exercise in patients with chronic thromboembolic pulmonary hypertension after balloon pulmonary angioplasty (THERAPY-HYBRID-BPA trial). BMJ Open. 2023 Jul 5;13(7):e072241. doi: 10.1136/bmjopen-2023-072241. PMID 37407055
- [Derived] Shimokawahara H, Ogawa A, Matsubara H. Balloon pulmonary angioplasty for chronic thromboembolic pulmonary hypertension: advances in patient and lesion selection. Curr Opin Pulm Med. 2021 Sep 1;27(5):303-310. doi: 10.1097/MCP.0000000000000797. PMID 34224432